CLINICAL TRIAL: NCT02949011
Title: A Phase 3, Multicenter, Randomized, Double-blind Study of a Single Dose of S-033188 Compared With Placebo or Oseltamivir 75 mg Twice Daily for 5 Days in Patients With Influenza at High Risk of Influenza Complications
Brief Title: Study of S-033188 (Baloxavir Marboxil) Compared With Placebo or Oseltamivir in Patients With Influenza at High Risk of Influenza Complications
Acronym: CAPSTONE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1602T0832; 2016-002688-32 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Results first posted 2019-11-06 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Influenza
Keywords: Tamiflu®; Influenza; Oseltamivir; Flu; S-033188
MeSH Terms: conditions — Influenza, Human | interventions — baloxavir; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Baloxavir Marboxil (Experimental): Participants received either 40 mg or 80 mg of baloxavir marboxil orally on Day 1 based on body weight of < 80 kg or ≥ 80 kg at Screening, respectively. Participants also received placebo to oseltamivir orally twice a day (BID) on Days 1 to 5.
  Interventions: Drug: Baloxavir Marboxil; Drug: Placebo to Oseltamivir
- Oseltamivir (Active Comparator): Participants received 75 mg oseltamivir twice a day on Days 1 to 5 and placebo to baloxavir marboxil on Day 1.
  Interventions: Drug: Placebo to Baloxavir Marboxil; Drug: Oseltamivir
- Placebo (Placebo Comparator): Participants received placebo to baloxavir marboxil on Day 1 and placebo to oseltamivir orally twice a day on Days 1 to 5.
  Interventions: Drug: Placebo to Baloxavir Marboxil; Drug: Placebo to Oseltamivir

INTERVENTIONS:
Drug: Baloxavir Marboxil — Tablets taken orally
  Other Names: S-033188; Xofluza®
  Arms: Baloxavir Marboxil
Drug: Placebo to Baloxavir Marboxil — Matching tablets taken orally
  Arms: Oseltamivir; Placebo
Drug: Oseltamivir — Capsules taken orally
  Other Names: Tamiflu®
  Arms: Oseltamivir
Drug: Placebo to Oseltamivir — Matching placebo capsules taken orally
  Arms: Baloxavir Marboxil; Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy of a single, oral dose of baloxavir marboxil compared with placebo by measuring the time to improvement of influenza symptoms in patients with influenza presenting within 48 hours of symptom onset.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians who provide written informed consent to participate in the study on a voluntary basis. For adolescent patients, informed consent/assent of voluntary participation should be obtained in accordance with local requirements.
2. Male or female patients ≥ 12 years at the time of signing the informed consent/assent form.
3. Patients with a diagnosis of influenza confirmed by all of the following:

   1. Fever ≥ 38ºC (axillary) during the predose examinations or within the 4 hours prior if antipyretics were taken
   2. A positive rapid influenza diagnostic test (RIDT) result OR A patient with a negative RIDT may be enrolled if the patient reports contact with a known case of influenza within the prior 7 days and all other inclusion criteria are met.
   3. At least 1 each of the following general and respiratory symptoms associated with influenza is present with a severity of moderate or greater:

   i. General symptoms (headache, feverishness or chills, muscle or joint pain, or fatigue) ii. Respiratory symptoms (cough, sore throat, or nasal congestion)
4. The time interval between the onset of symptoms and the predose examinations is 48 hours or less. The onset of symptoms is defined as either:

   1. Time of the first increase in body temperature (an increase of at least 1ºC from normal body temperature)
   2. Time when the patient experiences at least 1 new general or respiratory symptom
5. If a women of childbearing potential, agrees to use a highly effective method of contraception for 3 months after the first dose of study drug
6. Patients will be considered at high risk* of influenza complications due to the presence of at least 1 of the following inclusion criteria:

   1. Asthma or chronic lung disease (such as chronic obstructive pulmonary disease or cystic fibrosis)
   2. Endocrine disorders (including diabetes mellitus)
   3. Residents of long-term care facilities (eg, nursing homes)
   4. Compromised immune system (including patients receiving corticosteroids not exceeding 20 mg of prednisolone or equivalent, and patients being treated for human immunodeficiency virus [HIV] infection with a CD4 count > 350 cells/mm³ within the last 6 months)
   5. Neurological and neurodevelopmental disorders (including disorders of the brain, spinal cord, peripheral nerve, and muscle, eg, cerebral palsy, epilepsy [seizure disorders], stroke, muscular dystrophy, or spinal cord injury)
   6. Heart disease (such as congenital heart disease, congestive heart failure, or coronary artery disease), excluding hypertension without any other heart-related symptoms
   7. Adults aged ≥ 65 years
   8. American Indians and Alaskan Natives
   9. Blood disorders (such as sickle cell disease)
   10. Metabolic disorders (such as inherited metabolic disorders and mitochondrial disorders)
   11. Morbid obesity (body mass index ≥ 40 kg/m²)
   12. Women who are within 2 weeks postpartum and are not breastfeeding

Exclusion Criteria:

1. Patients with severe influenza virus infection requiring inpatient treatment.
2. Patients with known allergy to oseltamivir (Tamiflu®).
3. Patients unable to swallow tablets or capsules.
4. Patients who have previously received baloxavir marboxil.
5. Patients weighing ≤ 40 kg.
6. Patients who have been exposed to an investigational drug within 30 days prior to the predose examinations.
7. Women who are pregnant, breastfeeding, or have a positive pregnancy test at the predose examinations. The following female patients who have documentation of either a or b below do not need to undergo a pregnancy test at the predose examinations:

   1. Postmenopausal women (defined as cessation of regular menstrual periods for 2 years or more and confirmed by a follicle-stimulating hormone test)
   2. Women who are surgically sterile by hysterectomy, bilateral oophorectomy, or tubal ligation
8. Patients with concurrent infections at the predose examinations requiring systemic antimicrobial therapy.
9. Patients with liver disease associated with hepatic impairment.
10. Patients with cancer within the last 5 years (unless nonmelanoma skin cancer).
11. Patients with untreated HIV infection or treated HIV infection with a CD4 count below 350 cells/mm3 in the last 6 months.
12. Patients with immunosuppression following organ or bone marrow transplants.
13. Patients exceeding 20 mg of prednisolone or equivalent dose of chronic systemic corticosteroids.
14. Patients who have received peramivir, laninamivir, oseltamivir, zanamivir, rimantadine, umifenovir or amantadine within 30 days prior to the predose examinations.
15. Patients who have received an investigational monoclonal antibody for a viral disease in the last year.
16. Patients with known creatinine clearance ≤ 60 mL/min.
17. Patients who, in the opinion of the investigator, would be unlikely to comply with required study visits, self-assessments, and interventions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2184 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi

REFERENCES:
- [Derived] Retout S, De Buck S, Jolivet S, Duval V, Cosson V. A Pharmacokinetics-Time to Alleviation of Symptoms Model to Support Extrapolation of Baloxavir Marboxil Clinical Efficacy in Different Ethnic Groups with Influenza A or B. Clin Pharmacol Ther. 2022 Aug;112(2):372-381. doi: 10.1002/cpt.2648. Epub 2022 Jun 10. PMID 35585696
- [Derived] Ison MG, Portsmouth S, Yoshida Y, Shishido T, Mitchener M, Tsuchiya K, Uehara T, Hayden FG. Early treatment with baloxavir marboxil in high-risk adolescent and adult outpatients with uncomplicated influenza (CAPSTONE-2): a randomised, placebo-controlled, phase 3 trial. Lancet Infect Dis. 2020 Oct;20(10):1204-1214. doi: 10.1016/S1473-3099(20)30004-9. Epub 2020 Jun 8. PMID 32526195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 551 sites, including 242 sites in the United States, 142 sites in Japan, 48 sites in APAC (including Australia, New Zealand, Philippines, and South Korea), 98 sites in Europe (Belgium, Germany, Hungary, Latvia, Poland, Romania, and Spain), and 21 sites in South Africa.
Pre-assignment Details: Eligible patients were randomized in a 1:1:1 ratio to 1 of 3 treatment groups. Participants were stratified by baseline symptom score (≤ 14 or ≥ 15), preexisting and worsened symptom (Yes or No), region (Asia, North America/Europe, or Southern Hemisphere), and patient's weight (< 80 kg or ≥ 80 kg).
Period: Overall Study
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Started | 730 | 729 | 725
Received Study Drug | 728 | 728 (Includes one participant who received baloxavir marboxil in error) | 722 (Includes one participant who received baloxavir marboxil in error)
Intention to Treat Infected Population | 388 | 386 | 389
Completed | 697 | 695 | 683
Not Completed | 33 | 34 | 42
Not completed — Adverse Event | 6 | 7 | 3
Not completed — Failed Inclusion/Exclusion Criteria | 0 | 0 | 3
Not completed — Protocol Deviation | 5 | 3 | 3
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Withdrawal by Subject | 13 | 13 | 21
Not completed — Lost to Follow-up | 7 | 5 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Miscellaneous | 2 | 4 | 6

BASELINE CHARACTERISTICS:
Population: The Intention-to-treat Infected population includes all participants with a confirmed diagnosis of influenza virus infection who received study drug, and were enrolled at sites with Good Clinical Practice compliance. Confirmation of influenza virus infection was based on the results of reverse transcription polymerase chain reaction on Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir | Total
Number analyzed (Participants) | 388 | 386 | 389 | 1163
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (16.8) | 51.9 (16.7) | 51.1 (17.0) | 51.8 (16.8)
Age, Customized [Count of Participants; unit: Participants]
  ≥ 12 to ≤ 19 years | 19 | 17 | 22 | 58
  ≥ 20 to ≤ 29 years | 29 | 22 | 27 | 78
  ≥ 30 to ≤ 39 years | 42 | 58 | 44 | 144
  ≥ 40 to ≤ 49 years | 63 | 55 | 75 | 193
  ≥ 50 to ≤ 59 years | 83 | 101 | 83 | 267
  ≥ 60 to ≤ 64 years | 39 | 30 | 35 | 104
  ≥ 65 to ≤ 74 years | 85 | 76 | 78 | 239
  ≥ 75 years | 28 | 27 | 25 | 80
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 206 | 198 | 599
  Male | 193 | 180 | 191 | 564
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 59 | 56 | 177
  Not Hispanic or Latino | 325 | 327 | 331 | 983
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3 | 6
  Asian | 167 | 157 | 163 | 487
  Black or African American | 39 | 30 | 29 | 98
  White | 178 | 194 | 188 | 560
  Other | 3 | 3 | 6 | 12
Weight [Count of Participants; unit: Participants]
  < 80 kg | 239 | 232 | 233 | 704
  ≥ 80 kg | 149 | 154 | 156 | 459
Time to Treatment From Influenza Onset [Count of Participants; unit: Participants]
  ≥ 0 to ≤ 12 hours | 27 | 42 | 37 | 106
  > 12 to ≤ 24 hours | 151 | 150 | 119 | 420
  > 24 to ≤ 36 hours | 114 | 120 | 141 | 375
  > 36 to ≤ 48 hours | 95 | 74 | 92 | 261
  Missing | 1 | 0 | 0 | 1
Influenza Virus Subtype Based on RT-PCR Assay [Count of Participants; unit: Participants]
  A/H1N1pdm | 28 | 17 | 35 | 80
  A/H3 | 182 | 185 | 190 | 557
  B | 167 | 168 | 149 | 484
  Mixed infection | 4 | 5 | 5 | 14
  Other | 7 | 11 | 10 | 28
Influenza Virus Titer [Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]] — Virus titer was quantified from nasopharyngeal swabs (or throat swabs if nasopharyngeal swabbing was not feasible) by tissue culture methods. Population: Participants with available virus titer data
  log₁₀[TCID₅₀/mL]
    number analyzed (Participants) | 378 | 377 | 380 | 1135
    (all) | 4.96 (2.28) | 5.27 (2.39) | 5.25 (2.27) | 5.16 (2.32)
Influenza Virus Ribonucleic Acid (RNA) Load [Mean (Standard Deviation); unit: log₁₀ virus particles/mL] — Virus RNA was measured by reverse transcription polymerase chain reaction (RT-PCR) from nasopharyngeal swabs (or throat swabs, if nasopharyngeal swabbing was not feasible. Population: Participants with available influenza virus RNA data
  log₁₀ virus particles/mL
    number analyzed (Participants) | 385 | 378 | 387 | 1150
    (all) | 6.72 (1.43) | 6.87 (1.54) | 6.81 (1.37) | 6.80 (1.45)
Region [Count of Participants; unit: Participants]
  Asia | 159 | 151 | 152 | 462
  North America/Europe | 212 | 216 | 220 | 648
  Southern Hemisphere | 17 | 19 | 17 | 53
Composite Symptom Score [Count of Participants; unit: Participants] — Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). The composite symptom score is the total score of the 7 influenza symptoms as assessed by the participant, and ranges from 0 to 21.
  Participants
    ≤ 14 | 188 | 188 | 201 | 577
    ≥ 15 | 200 | 198 | 188 | 586
Preexisting Symptom Status [Count of Participants; unit: Participants] — Preexisting symptoms include cough, fatigue, or muscle/joint pain that existed prior to developing influenza.
  Participants were asked at baseline if they had any of these preexisting symptoms in the past 30 days, and if they were worsened by the onset of influenza.
  Participants with at least 1 of the above 3 symptoms prior to onset of influenza that worsened with the onset of influenza were categorized as "Yes", and all other participants (preexisting symptoms but not worsened or no preexisting symptoms) were categorized as "No".
  Participants
    Yes | 71 | 76 | 69 | 216
    No | 317 | 310 | 320 | 947

OUTCOME MEASURES:

1. Primary Outcome: Time to Improvement of Influenza Symptoms
Description: Participants assessed the severity of 7 influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness/chills, muscle/joint pain, and fatigue) on a 4-point scale (0 = no symptoms, 1= mild, 2 = moderate, and 3 = severe). Time to improvement of symptoms was defined as the time from the start of treatment to the time when all influenza symptoms were alleviated, maintained, or improved, as defined below, for a duration of at least 21.5 hours:
  * Preexisting symptoms (cough, fatigue, or muscle/joint pain that existed prior to influenza) that were worse at baseline must have improved at least 1 point from baseline
  * Preexisting symptoms not worse at baseline must have maintained baseline severity
  * New symptoms must have alleviated, defined as a symptom score of none (0) or mild (1).
  Time to improvement of symptoms was analyzed using Kaplan-Meier (KM) methods; participants who did not experience improvement of symptom s were censored at the last observation.
Time Frame: From Day 1 pretreatment up to Day 14
Population: Participants in the intention-to-treat infected population with available time to improvement of symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 385 | 385 | 388
hours | 73.2 [67.2 to 85.1] | 102.3 [92.7 to 113.1] | 81.0 [69.4 to 91.5]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; The primary analysis of the primary endpoint was a comparison between the baloxavir marboxil and placebo groups; Test type: Superiority; p < 0.0001, Stratified generalized Wilcoxon test — Adjusted p-value, two-sided significance level of 0.05; Peto-Prentice's generalized Wilcoxon test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region; Median Difference = -29.1, 95% CI 2-sided [-42.8 to -14.6]
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; The comparison between the baloxavir marboxil and the oseltamivir groups was conducted as a secondary analysis only if a statistically significant difference was observed in the primary analysis in order to maintain control of overall type I error; Test type: Superiority; p = 0.8347, Stratified generalized Wilcoxon test — Adjusted p-value, two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -7.7, 95% CI 2-sided [-22.7 to 7.9]
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; Analysis using the stratified log rank test was performed as a sensitivity analysis; Test type: Superiority; p = 0.0008, Log Rank — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Log rank test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; Analysis using the stratified log rank test was performed as a sensitivity analysis; Test type: Superiority; p = 0.8449, Log Rank — The p-value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Log rank test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

2. Secondary Outcome: Percentage of Participants With Positive Influenza Virus Titer at Each Time Point
Description: Virus titer was quantified from nasopharyngeal swabs (or throat swabs if nasopharyngeal swabbing was not feasible) using tissue culture methods. Positive influenza virus titer was defined as virus titer not less than the lower limit of quantification (0.7 log₁₀ of the 50% tissue culture infective dose (TCID₅₀/mL) among those assessed for virus titer on Days 2, 3, 4, 5, 6, and 9.
Time Frame: Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infected population with a positive influenza virus titer on Day 1 and with available virus titer data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 355 | 353 | 360
percentage of participants
  Day 2: number analyzed (Participants) | 336 | 344 | 344
  Day 2 | 58.6 [53.2 to 63.9] | 86.9 [82.9 to 90.3] | 86.9 [82.9 to 90.3]
  Day 3: number analyzed (Participants) | 338 | 337 | 340
  Day 3 | 31.7 [26.7 to 36.9] | 72.7 [67.6 to 77.4] | 60.0 [54.6 to 65.2]
  Day 4: number analyzed (Participants) | 130 | 122 | 124
  Day 4 | 18.5 [12.2 to 26.2] | 50.0 [40.8 to 59.2] | 33.1 [24.9 to 42.1]
  Day 5: number analyzed (Participants) | 326 | 322 | 333
  Day 5 | 16.0 [12.1 to 20.4] | 30.7 [25.7 to 36.1] | 20.4 [16.2 to 25.2]
  Day 6: number analyzed (Participants) | 115 | 106 | 105
  Day 6 | 4.3 [1.4 to 9.9] | 16.0 [9.6 to 24.4] | 11.4 [6.0 to 19.1]
  Day 9: number analyzed (Participants) | 327 | 321 | 322
  Day 9 | 2.8 [1.3 to 5.2] | 5.3 [3.1 to 8.3] | 0.9 [0.2 to 2.7]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Day 2; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 2; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; Day 3; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 3; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; Day 4; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 4; Test type: Superiority; p = 0.0044, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; Day 5; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 5; Test type: Superiority; p = 0.1146, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; Day 6; Test type: Superiority; p = 0.0046, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 6; Test type: Superiority; p = 0.441, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; Day 9; Test type: Superiority; p = 0.0929, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 9; Test type: Superiority; p = 0.0907, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

3. Secondary Outcome: Percentage of Participants With Positive Influenza Virus by RT-PCR at Each Time Point
Description: Influenza virus ribonucleic acid (RNA) was quantified from nasopharyngeal swabs (or throat swabs, if nasopharyngeal swabbing was not feasible). The percentage of participants with detectable virus RNA (2.05 for flu A and 2.83 for flu B log₁₀ virus particles/mL) measured by reverse transcription polymerase chain reaction (RT-PCR) among those assessed on Days 2, 3, 4, 5, 6 and 9.
Time Frame: Days 2, 3, 4 (optional), 5, 6 (optional), and 9.
Population: Participants in the intention-to-treat infected population with positive influenza virus RNA determined by RT-PCR on Day 1 and with available data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 388 | 386 | 389
percentage of participants
  Day 2: number analyzed (Participants) | 371 | 375 | 374
  Day 2 | 96.0 [93.4 to 97.7] | 96.3 [93.8 to 97.9] | 96.0 [93.5 to 97.7]
  Day 3: number analyzed (Participants) | 375 | 372 | 369
  Day 3 | 92.5 [89.4 to 95.0] | 95.4 [92.8 to 97.3] | 95.1 [92.4 to 97.1]
  Day 4: number analyzed (Participants) | 148 | 144 | 140
  Day 4 | 86.5 [79.9 to 91.5] | 91.0 [85.1 to 95.1] | 86.4 [79.6 to 91.6]
  Day 5: number analyzed (Participants) | 364 | 361 | 361
  Day 5 | 84.9 [80.8 to 88.4] | 88.6 [84.9 to 91.7] | 86.1 [82.2 to 89.5]
  Day 6: number analyzed (Participants) | 131 | 123 | 117
  Day 6 | 71.8 [63.2 to 79.3] | 78.0 [69.7 to 85.0] | 71.8 [62.7 to 79.7]
  Day 9: number analyzed (Participants) | 363 | 356 | 350
  Day 9 | 54.5 [49.3 to 59.8] | 64.9 [59.7 to 69.8] | 57.7 [52.3 to 62.9]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Day 2; Test type: Superiority; p = 0.7383, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 2; Test type: Superiority; p = 0.9619, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; Day 3; Test type: Superiority; p = 0.0576, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 3; Test type: Superiority; p = 0.1237, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; Day 4; Test type: Superiority; p = 0.3071, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 4; Test type: Superiority; p = 0.9603, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; Day 5; Test type: Superiority; p = 0.0784, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 5; Test type: Superiority; p = 0.5547, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; Day 6; Test type: Superiority; p = 0.3087, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 6; Test type: Superiority; p = 0.9106, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; Day 9; Test type: Superiority; p = 0.0017, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 9; Test type: Superiority; p = 0.3068, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

4. Secondary Outcome: Change From Baseline in Virus Titer at Each Time Point
Description: Virus titer was quantified from nasopharyngeal swabs (or throat swabs if nasopharyngeal swabbing was not feasible) by tissue culture methods.
  If virus titer was less than the lower limit of quantification, the virus titer was imputed 0.7 (TCID₅₀/mL).
Time Frame: Day 1 pretreatment (Baseline) and Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infected population with positive influenza virus titer on Day 1 and with available virus titer data at each time point.
Measure: Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 355 | 353 | 360
log₁₀[TCID₅₀/mL]
  Day 2: number analyzed (Participants) | 336 | 343 | 344
  Day 2 | -3.36 (2.21) | -1.25 (2.27) | -1.76 (2.20)
  Day 3: number analyzed (Participants) | 338 | 336 | 340
  Day 3 | -3.92 (2.22) | -2.99 (2.55) | -3.26 (2.50)
  Day 4: number analyzed (Participants) | 130 | 121 | 124
  Day 4 | -3.99 (2.00) | -3.79 (2.75) | -3.75 (2.26)
  Day 5: number analyzed (Participants) | 326 | 321 | 333
  Day 5 | -4.32 (2.16) | -4.38 (2.31) | -4.41 (2.12)
  Day 6: number analyzed (Participants) | 115 | 105 | 105
  Day 6 | -4.07 (2.05) | -4.68 (2.22) | -4.39 (1.97)
  Day 9: number analyzed (Participants) | 327 | 320 | 322
  Day 9 | -4.53 (2.11) | -4.91 (2.08) | -4.78 (2.07)
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; Day 3; Test type: Superiority; p < 0.0001, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 3; Test type: Superiority; p = 0.0024, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; Day 4; Test type: Superiority; p = 0.9127, ven Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 4; Test type: Superiority; p = 0.5361, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; Day 5; Test type: Superiority; p = 0.5739, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 5; Test type: Superiority; p = 0.5466, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; Day 6; Test type: Superiority; p = 0.0543, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 6; Test type: Superiority; p = 0.4677, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; Day 9; Test type: Superiority; p = 0.0266, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 9; Test type: Superiority; p = 0.1281, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

5. Secondary Outcome: Change From Baseline in Virus RNA (RT-PCR) at Each Time Point
Description: Nasopharyngeal swabs (or throat swabs, if nasopharyngeal swabbing was not feasible) were obtained for viral quantitation. Virus RNA was measured by reverse transcription polymerase chain reaction (RT-PCR).
Time Frame: Day 1 pretreatment (Baseline) and Days 2, 3, 4 (optional), 5, 6 (optional), and 9
Population: Participants in the intention-to-treat infected population with positive RT-PCR on Day 1 and with available virus RNA data at each time point.
Measure: Mean (Standard Deviation); unit: log₁₀ virus particles/mL
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 388 | 386 | 389
log₁₀ virus particles/mL
  Day 2: number analyzed (Participants) | 369 | 370 | 373
  Day 2 | -1.13 (1.20) | -0.62 (1.34) | -0.76 (1.18)
  Day 3: number analyzed (Participants) | 374 | 366 | 368
  Day 3 | -2.09 (1.45) | -1.57 (1.66) | -1.77 (1.45)
  Day 4: number analyzed (Participants) | 147 | 138 | 139
  Day 4 | -2.77 (1.42) | -2.09 (1.84) | -2.34 (1.63)
  Day 5: number analyzed (Participants) | 361 | 353 | 359
  Day 5 | -3.09 (1.58) | -2.77 (1.67) | -3.04 (1.46)
  Day 6: number analyzed (Participants) | 129 | 119 | 116
  Day 6 | -3.33 (1.48) | -3.19 (1.77) | -3.41 (1.38)
  Day 9: number analyzed (Participants) | 360 | 349 | 349
  Day 9 | -3.89 (1.51) | -3.78 (1.65) | -3.99 (1.39)
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 2; Test type: Superiority; p < 0.0001, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; Day 3; Test type: Superiority; p < 0.0001, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 3; Test type: Superiority; p = 0.0015, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; Day 4; Test type: Superiority; p = 0.0028, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 4; Test type: Superiority; p = 0.0265, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; Day 5; Test type: Superiority; p = 0.0247, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 5; Test type: Superiority; p = 0.5298, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; Day 6; Test type: Superiority; p = 0.9554, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 6; Test type: Superiority; p = 0.9075, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; Day 9; Test type: Superiority; p = 0.7624, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; Day 9; Test type: Superiority; p = 0.6156, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

6. Secondary Outcome: Area Under the Curve (AUC) Adjusted by Baseline in Influenza Virus Titer
Description: This endpoint was defined as AUC of change from Baseline in virus titer from Day 1 to Day 9. AUC was calculated using the trapezoidal method.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infected population with a positive virus titer on Day 1 and available sample on Day 9.
Measure: Mean (Standard Deviation); unit: log₁₀[TCID₅₀/mL]*hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 355 | 353 | 360
log₁₀[TCID₅₀/mL]*hours | -727.7 (367.2) | -660.2 (372.3) | -695.5 (360.5)
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.0340, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.2766, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

7. Secondary Outcome: Area Under the Curve (AUC) Adjusted by Baseline in Viral RNA
Description: This endpoint was defined as AUC of change from baseline in the amount of virus RNA (RT-PCR) from Day 1 to Day 9. The AUC was calculated using the trapezoidal method.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infected population with a positive virus RNA determined by RT-PCR at baseline and available sample on Day 9.
Measure: Mean (Standard Deviation); unit: log₁₀ virus particles/mL*hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 360 | 349 | 349
log₁₀ virus particles/mL*hours | -490.9 (249.3) | -434.9 (269.3) | -482.2 (233.2)
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.0072, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.7330, van Elteren test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Van Elteren test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

8. Secondary Outcome: Time to Cessation of Viral Shedding Determined by Virus Titer
Description: Time to cessation of viral shedding by virus titer was defined as the time between the initiation of the study treatment and first time when the virus titer was below the limit of detection (0.7 log₁₀[TCID₅₀/mL]). The median and 95% confidence interval (CI) for time to cessation of viral shedding determined by virus titer was analyzed using the Kaplan-Meier (KM) method; participants whose virus titer had not reached cessation by the last observation time point were treated as censored at that time point.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infected population with a positive virus titer on Day 1 whose time to cessation of viral shedding by virus titer was not missing.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 352 | 352 | 356
hours | 48.0 [NA to NA] — Could not be estimated because lower limit of 95% CI of KM survival function just before the median survival time was higher than 50% and an upper limit of 95% CI of KM survival function just after the median survival time was lower than 50%. | 96.0 [NA to NA] — Could not be estimated because lower limit of 95% CI of KM survival function just before the median survival time was higher than 50% and an upper limit of 95% CI of KM survival function just after the median survival time was lower than 50%. | 96.0 [72.0 to 96.0]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -48.0, 95% CI 2-sided [-48.0 to -48.0]
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -48.0, 95% CI 2-sided [-48.0 to -24.0]

9. Secondary Outcome: Time to Cessation of Viral Shedding Determined by Virus RNA
Description: Time to cessation of viral shedding by RT-PCR was defined as the time between the initiation of the study treatment and first time when the virus RNA was below the limit of detection measured by RT-PCR.
  Time to cessation of viral shedding by RT-PCR was analyzed using the KM method; participants whose virus RNA had not reached cessation by the last observation time point were treated as censored at that time point.
Time Frame: Day 1 to Day 9
Population: Participants in the intention-to-treat infected population with positive influenza virus RNA determined by RT-PCR on Day 1 whose time to cessation of viral shedding by RT-PCR.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 385 | 385 | 384
hours | 216.0 [192.0 to 240.0] | 240.0 [216.0 to 312.0] | 216.0 [216.0 to 240.0]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.0006, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -24.0, 95% CI 2-sided [-96.0 to 0.0]
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.2370, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = 0.0, 95% CI 2-sided [-48.0 to 24.0]

10. Secondary Outcome: Percentage of Participants Whose Symptoms Were Improved at Each Time Point
Description: Participants assessed the severity of 7 influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (0 = no symptoms, 1= mild, 2 = moderate, and 3 = severe).
  Improvement of symptoms was defined as all influenza symptoms alleviated, maintained, or improved, as defined below, for a duration of at least 21.5 hours:
  * Preexisting symptoms (cough, fatigue, or muscle/joint pain that existed prior to influenza) judged to be worse at baseline must have improved at least 1 point from baseline severity
  * Preexisting symptoms judged not to be worse at baseline must have maintained baseline severity
  * New symptoms at baseline must have alleviated, defined as a symptom score of none (0) or mild (1).
Time Frame: 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, and 216 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infected population with available symptoms data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 388 | 386 | 389
percentage of participants
  12 hours: number analyzed (Participants) | 297 | 303 | 307
  12 hours | 9.1 [6.1 to 13.0] | 8.6 [5.7 to 12.3] | 8.1 [5.3 to 11.8]
  24 hours: number analyzed (Participants) | 357 | 365 | 367
  24 hours | 18.8 [14.9 to 23.2] | 14.2 [10.8 to 18.3] | 19.6 [15.7 to 24.1]
  36 hours: number analyzed (Participants) | 304 | 304 | 300
  36 hours | 33.9 [28.6 to 39.5] | 21.1 [16.6 to 26.1] | 31.0 [25.8 to 36.6]
  48 hours: number analyzed (Participants) | 363 | 368 | 363
  48 hours | 38.0 [33.0 to 43.2] | 28.8 [24.2 to 33.7] | 39.9 [34.9 to 45.2]
  72 hours: number analyzed (Participants) | 359 | 359 | 350
  72 hours | 56.0 [50.7 to 61.2] | 41.8 [36.6 to 47.1] | 56.0 [50.6 to 61.3]
  96 hours: number analyzed (Participants) | 352 | 341 | 350
  96 hours | 65.9 [60.7 to 70.9] | 53.4 [47.9 to 58.8] | 61.1 [55.8 to 66.3]
  120 hours: number analyzed (Participants) | 358 | 342 | 333
  120 hours | 72.3 [67.4 to 76.9] | 64.6 [59.3 to 69.7] | 72.4 [67.2 to 77.1]
  144 hours: number analyzed (Participants) | 347 | 342 | 330
  144 hours | 78.1 [73.4 to 82.3] | 69.6 [64.4 to 74.4] | 77.6 [72.7 to 82.0]
  168 hours: number analyzed (Participants) | 342 | 326 | 333
  168 hours | 80.1 [75.5 to 84.2] | 72.7 [67.5 to 77.5] | 79.6 [74.8 to 83.8]
  192 hours: number analyzed (Participants) | 341 | 337 | 327
  192 hours | 83.6 [79.2 to 87.3] | 78.0 [73.2 to 82.3] | 85.6 [81.3 to 89.2]
  216 hours: number analyzed (Participants) | 197 | 174 | 178
  216 hours | 85.8 [80.1 to 90.3] | 78.7 [71.9 to 84.6] | 88.2 [82.5 to 92.5]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; 12 hours; Test type: Superiority; p = 0.7698, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; 12 hours; Test type: Superiority; p = 0.5777, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; 24 hours; Test type: Superiority; p = 0.1112, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; 24 hours; Test type: Superiority; p = 0.6483, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; 36 hours; Test type: Superiority; p = 0.0004, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; 36 hours; Test type: Superiority; p = 0.5625, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; 48 hours; Test type: Superiority; p = 0.0072, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; 48 hours; Test type: Superiority; p = 0.6234, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; 72 hours; Test type: Superiority; p = 0.0002, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; 72 hours; Test type: Superiority; p = 0.9547, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; 96 hours; Test type: Superiority; p = 0.0012, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; 96 hours; Test type: Superiority; p = 0.1860, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 13: Comparison: Baloxavir Marboxil vs Placebo; 120 hours; Test type: Superiority; p = 0.0274, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 14: Comparison: Baloxavir Marboxil vs Oseltamivir; 120 hours; Test type: Superiority; p = 0.9635, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 15: Comparison: Baloxavir Marboxil vs Placebo; 144 hours; Test type: Superiority; p = 0.0081, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 16: Comparison: Baloxavir Marboxil vs Oseltamivir; 144 hours; Test type: Superiority; p = 0.7425, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 17: Comparison: Baloxavir Marboxil vs Placebo; 168 hours; Test type: Superiority; p = 0.0209, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 18: Comparison: Baloxavir Marboxil vs Oseltamivir; 168 hours; Test type: Superiority; p = 0.7448, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 19: Comparison: Baloxavir Marboxil vs Placebo; 192 hours; Test type: Superiority; p = 0.0644, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 20: Comparison: Baloxavir Marboxil vs Oseltamivir; 192 hours; Test type: Superiority; p = 0.4931, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 21: Comparison: Baloxavir Marboxil vs Placebo; 216 hours; Test type: Superiority; p = 0.0708, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 22: Comparison: Baloxavir Marboxil vs Oseltamivir; 216 hours; Test type: Superiority; p = 0.4024, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel-Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

11. Secondary Outcome: Time to Alleviation of Symptoms
Description: Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of symptoms was defined as the time from the start of the study treatment to the time when all seven influenza-related symptoms were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours.
  Time to alleviation of symptoms was analyzed using Kaplan-Meier (KM) methods; participants who did not experience alleviation of symptoms were censored at the last observation time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infected population with available time to alleviation of symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 385 | 385 | 388
hours | 77.0 [68.4 to 88.3] | 102.8 [93.2 to 113.4] | 85.6 [71.5 to 94.8]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -25.8
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.9127, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -8.6

12. Secondary Outcome: Time to Improvement of the Four Systemic Symptoms
Description: Participants assessed the severity of 7 influenza-associated symptoms on a 4-point scale (from 0 = no symptoms to 3 = severe symptoms). Time to improvement of the 4 systemic symptoms was defined as the time between the initiation of study treatment to the time when all 4 systemic symptoms (headache, feverishness or chills, muscle or joint pain, and fatigue) were alleviated, maintained, or improved, as defined below, for a duration of at least 21.5 hours:
  * Preexisting symptoms (cough, fatigue, or muscle/joint pain that existed prior to influenza) that were worse at baseline must have improved at least 1 point from baseline
  * Preexisting symptoms not worse at baseline must have maintained baseline severity
  * New symptoms at baseline must have alleviated, defined as a symptom score of none (0) or mild (1).
  Time to improvement of the 4 systemic symptoms was analyzed using KM methods; participants who did not experience improvement of symptoms were censored at the last observation.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infected population with available time to improvement of the 4 systemic symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 385 | 385 | 388
hours | 51.7 [45.0 to 55.4] | 66.8 [60.1 to 70.0] | 49.4 [44.2 to 56.8]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.0013, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -15.1
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.8498, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = 2.3

13. Secondary Outcome: Time to Improvement of the Three Respiratory Symptoms
Description: Participants assessed the severity of 7 influenza-associated symptoms on a 4-point scale (from 0 = no symptoms to 3 = severe symptoms). Time to improvement of the 3 respiratory symptoms was defined as the time from the start of study treatment to the time when all 3 respiratory symptoms (cough, sore throat, and nasal congestion) were alleviated, maintained, or improved, as defined below, for a duration of at least 21.5 hours:
  * Preexisting symptoms (cough, fatigue, or muscle/joint pain that existed prior to influenza) that were worse at baseline must have improved at least 1 point from baseline
  * Preexisting symptoms not worse at baseline must have maintained baseline severity
  * New symptoms at baseline must have alleviated, defined as a symptom score of none (0) or mild (1).
  Time to improvement of the 3 respiratory symptoms was analyzed using KM methods; participants who did not experience improvement of symptoms were censored at the last observation time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infected population with available time to improvement of the 3 respiratory symptoms data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 385 | 385 | 388
hours | 63.6 [55.9 to 68.2] | 87.8 [76.3 to 98.9] | 62.1 [54.0 to 69.1]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.0001, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -24.1
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.9237, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = 1.5

14. Secondary Outcome: Time to Resolution of Fever
Description: Time to resolution of fever was defined as the time between the initiation of the study treatment and the resolution of fever. The resolution of fever was defined as the time when the participant's self-measured axillary temperature became less than 37ºC and was maintained at less than 37ºC for at least 12 hours. Time to resolution of fever was analyzed using KM methods; participants who did not experience resolution of fever by the last observation time point were censored at that time point.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infected population whose body temperature at baseline was more than 37°C and time to resolution of fever was not missing
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 380 | 385 | 383
hours | 30.8 [28.2 to 35.4] | 50.7 [44.6 to 58.8] | 34.3 [30.0 to 38.9]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p < 0.0001, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -19.8, 95% CI 2-sided [-28.8 to -12.5]
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.2425, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -3.5, 95% CI 2-sided [-9.1 to 2.7]

15. Secondary Outcome: Percentage of Participants Reporting Normal Temperature at Each Time Point
Description: Defined as the percentage of patrticipants whose axillary body temperature dropped to less than 37ºC after the initiation of the study treatment.
Time Frame: 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, and 216 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infected population whose body temperature at baseline was more than 37°C and with available body temperature data at each time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 385 | 386 | 386
percentage of participants
  12 hours: number analyzed (Participants) | 343 | 338 | 344
  12 hours | 29.7 [24.9 to 34.9] | 24.6 [20.1 to 29.5] | 25.9 [21.3 to 30.8]
  24 hours: number analyzed (Participants) | 360 | 370 | 368
  24 hours | 51.1 [45.8 to 56.4] | 43.2 [38.1 to 48.5] | 54.3 [49.1 to 59.5]
  36 hours: number analyzed (Participants) | 345 | 352 | 340
  36 hours | 68.1 [62.9 to 73.0] | 47.4 [42.1 to 52.8] | 64.1 [58.8 to 69.2]
  48 hours: number analyzed (Participants) | 367 | 371 | 360
  48 hours | 77.4 [72.8 to 81.6] | 59.3 [54.1 to 64.3] | 76.4 [71.7 to 80.7]
  72 hours: number analyzed (Participants) | 337 | 336 | 322
  72 hours | 84.0 [79.6 to 87.7] | 71.7 [66.6 to 76.5] | 82.6 [78.0 to 86.6]
  96 hours: number analyzed (Participants) | 337 | 331 | 318
  96 hours | 87.5 [83.5 to 90.9] | 79.8 [75.0 to 84.0] | 85.8 [81.5 to 89.5]
  120 hours: number analyzed (Participants) | 327 | 328 | 310
  120 hours | 86.2 [82.0 to 89.8] | 86.6 [82.4 to 90.1] | 88.4 [84.3 to 91.7]
  144 hours: number analyzed (Participants) | 319 | 324 | 302
  144 hours | 90.0 [86.1 to 93.0] | 86.1 [81.9 to 89.7] | 87.4 [83.1 to 90.9]
  168 hours: number analyzed (Participants) | 321 | 311 | 300
  168 hours | 87.9 [83.8 to 91.2] | 88.1 [84.0 to 91.5] | 87.7 [83.4 to 91.2]
  192 hours: number analyzed (Participants) | 317 | 312 | 294
  192 hours | 89.0 [85.0 to 92.2] | 87.5 [83.3 to 91.0] | 90.5 [86.5 to 93.6]
  216 hours: number analyzed (Participants) | 311 | 298 | 309
  216 hours | 89.1 [85.1 to 92.3] | 89.9 [85.9 to 93.1] | 89.6 [85.7 to 92.8]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; 12 hours; Test type: Superiority; p = 0.1713, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; 12 hours; Test type: Superiority; p = 0.2249, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; 24 hours; Test type: Superiority; p = 0.0387, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; 24 hours; Test type: Superiority; p = 0.3915, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; 36 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; 36 hours; Test type: Superiority; p = 0.2617, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; 48 hours; Test type: Superiority; p < 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; 48 hours; Test type: Superiority; p = 0.8808, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; 72 hours; Test type: Superiority; p = 0.0001, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; 72 hours; Test type: Superiority; p = 0.5923, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; 96 hours; Test type: Superiority; p = 0.0064, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; 96 hours; Test type: Superiority; p = 0.6746, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 13: Comparison: Baloxavir Marboxil vs Placebo; 120 hours; Test type: Superiority; p = 0.8167, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 14: Comparison: Baloxavir Marboxil vs Oseltamivir; 120 hours; Test type: Superiority; p = 0.3773, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 15: Comparison: Baloxavir Marboxil vs Placebo; 144 hours; Test type: Superiority; p = 0.1041, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 16: Comparison: Baloxavir Marboxil vs Oseltamivir; 144 hours; Test type: Superiority; p = 0.3328, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 17: Comparison: Baloxavir Marboxil vs Placebo; 168 hours; Test type: Superiority; p = 0.7867, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 18: Comparison: Baloxavir Marboxil vs Oseltamivir; 168 hours; Test type: Superiority; p = 0.8640, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 19: Comparison: Baloxavir Marboxil vs Placebo; 192 hours; Test type: Superiority; p = 0.6465, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 20: Comparison: Baloxavir Marboxil vs Oseltamivir; 192 hours; Test type: Superiority; p = 0.4265, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 21: Comparison: Baloxavir Marboxil vs Placebo; 216 hours; Test type: Superiority; p = 0.6568, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region
Statistical Analysis 22: Comparison: Baloxavir Marboxil vs Oseltamivir; 216 hours; Test type: Superiority; p = 0.6102, Mantel Haenszel — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; Mantel Haenszel test stratified by baseline composite symptom score, preexisting and worsened symptoms, and region

16. Secondary Outcome: Body Temperature at Each Time Point
Description: Participant's self-measured axillary temperature using an electronic thermometer.
Time Frame: 12, 24, 36, 48, 72, 96 and 120 hours after the initial dose of study treatment
Population: Participants in the intention-to-treat infected population with available temperature data at each time point.
Measure: Least Squares Mean (Standard Error); unit: °C
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 388 | 386 | 389
°C
  12 hours: number analyzed (Participants) | 344 | 338 | 344
  12 hours | 37.39 (0.07) | 37.53 (0.07) | 37.43 (0.07)
  24 hours: number analyzed (Participants) | 361 | 370 | 368
  24 hours | 36.84 (0.06) | 37.02 (0.06) | 36.80 (0.06)
  36 hours: number analyzed (Participants) | 346 | 352 | 340
  36 hours | 36.58 (0.06) | 36.94 (0.06) | 36.62 (0.06)
  48 hours: number analyzed (Participants) | 368 | 371 | 360
  48 hours | 36.44 (0.06) | 36.77 (0.06) | 36.50 (0.06)
  72 hours: number analyzed (Participants) | 338 | 336 | 322
  72 hours | 36.30 (0.05) | 36.46 (0.05) | 36.29 (0.05)
  96 hours: number analyzed (Participants) | 338 | 331 | 318
  96 hours | 36.26 (0.05) | 36.35 (0.05) | 36.24 (0.05)
  120 hours: number analyzed (Participants) | 328 | 328 | 310
  120 hours | 36.26 (0.05) | 36.27 (0.05) | 36.21 (0.05)
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; 12 hours; Test type: Superiority; p = 0.0408, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; ANCOVA with baseline composite symptom score, preexisting and worsened symptom, region, and body temperature at baseline as covariates; LS Mean Difference = -0.14, 95% CI 2-sided [-0.28 to -0.01], Standard Error of Mean 0.07
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; 12 hours; Test type: Superiority; p = 0.5324, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.04, 95% CI 2-sided [-0.18 to 0.09], Standard Error of Mean 0.07
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; 24 hours; Test type: Superiority; p = 0.0025, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.18, 95% CI 2-sided [-0.30 to -0.06], Standard Error of Mean 0.06
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; 24 hours; Test type: Superiority; p = 0.4874, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = 0.04, 95% CI 2-sided [-0.08 to 0.16], Standard Error of Mean 0.06
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; 36 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.36, 95% CI 2-sided [-0.47 to -0.24], Standard Error of Mean 0.06
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; 36 hours; Test type: Superiority; p = 0.5414, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.04, 95% CI 2-sided [-0.15 to 0.08], Standard Error of Mean 0.06
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; 48 hours; Test type: Superiority; p < 0.0001, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.33, 95% CI 2-sided [-0.44 to -0.22], Standard Error of Mean 0.06
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; 48 hours; Test type: Superiority; p = 0.3185, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.06, 95% CI 2-sided [-0.17 to 0.05], Standard Error of Mean 0.06
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; 72 hours; Test type: Superiority; p = 0.0025, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.16, 95% CI 2-sided [-0.26 to -0.06], Standard Error of Mean 0.05
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; 72 hours; Test type: Superiority; p = 0.8299, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = 0.01, 95% CI 2-sided [-0.09 to 0.11], Standard Error of Mean 0.05
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; 96 hours; Test type: Superiority; p = 0.0878, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.09, 95% CI 2-sided [-0.19 to 0.01], Standard Error of Mean 0.05
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; 96 hours; Test type: Superiority; p = 0.7498, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = 0.02, 95% CI 2-sided [-0.09 to 0.12], Standard Error of Mean 0.05
Statistical Analysis 13: Comparison: Baloxavir Marboxil vs Placebo; 120 hours; Test type: Superiority; p = 0.8030, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = -0.01, 95% CI 2-sided [-0.11 to 0.09], Standard Error of Mean 0.05
Statistical Analysis 14: Comparison: Baloxavir Marboxil vs Oseltamivir; 120 hours; Test type: Superiority; p = 0.3577, ANCOVA — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 16, analysis 1]; LS Mean Difference = 0.05, 95% CI 2-sided [-0.05 to 0.15], Standard Error of Mean 0.05

17. Secondary Outcome: Time to Improvement of Individual Symptoms
Description: Participants assessed the severity of 7 influenza-associated symptoms on a 4-point scale (0 = no symptoms to 3 = severe). Time to improvement of cough, fatigue, and muscle/joint pain was defined as the time from the start of treatment to the time when each symptom was alleviated, maintained, or improved, as defined below, for at least 21.5 hours:
  * Preexisting symptoms that were worse at baseline must have improved at least 1 point from baseline
  * Preexisting symptoms not worse at baseline must have maintained baseline severity
  * New symptoms must have alleviated, defined as a score of 0 (None) or 1 (Mild). Time to improvement of sore throat, headache, nasal congestion, and feverish/chills was defined as the time from the start of treatment to the time when the symptom was assessed as 0 (None) or 1 (Mild) for at least 21.5 hours.
  Time to improvement of symptoms was analyzed using KM methods; participants with no improvement of symptoms were censored at the last observation.
Time Frame: Initiation of study treatment up to Day 14
Population: Participants in the intention-to-treat infected population; the analysis of each individual symptom includes participants with new or preexisting and worsened symptom scores of moderate (2) or severe (3) at baseline, and with available time to improvement of symptom data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 388 | 386 | 389
hours
  Cough: number analyzed (Participants) | 314 | 312 | 317
  Cough | 47.3 [42.8 to 52.7] | 70.4 [56.5 to 79.5] | 47.5 [43.0 to 55.4]
  Sore Throat: number analyzed (Participants) | 249 | 243 | 226
  Sore Throat | 40.2 [32.4 to 46.1] | 46.5 [39.0 to 53.5] | 39.3 [30.1 to 42.8]
  Headache: number analyzed (Participants) | 251 | 258 | 266
  Headache | 33.4 [29.1 to 40.5] | 43.9 [33.6 to 46.2] | 31.3 [28.6 to 37.0]
  Nasal Congestion: number analyzed (Participants) | 240 | 267 | 257
  Nasal Congestion | 45.6 [37.4 to 54.3] | 57.7 [48.7 to 67.8] | 44.0 [36.4 to 50.3]
  Feverishness or Chills: number analyzed (Participants) | 348 | 347 | 347
  Feverishness or Chills | 28.3 [24.2 to 31.8] | 31.9 [28.6 to 41.2] | 29.1 [25.2 to 30.8]
  Muscle or Joint Pain: number analyzed (Participants) | 311 | 302 | 312
  Muscle or Joint Pain | 37.2 [31.5 to 41.6] | 44.9 [42.2 to 52.0] | 33.2 [30.2 to 39.5]
  Fatigue: number analyzed (Participants) | 332 | 330 | 325
  Fatigue | 41.3 [35.2 to 46.1] | 48.8 [42.7 to 55.4] | 43.2 [39.3 to 47.4]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Cough; Test type: Superiority; p = 0.0009, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -23.1
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Cough; Test type: Superiority; p = 0.4074, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -0.2
Statistical Analysis 3: Comparison: Baloxavir Marboxil vs Placebo; Sore Throat; Test type: Superiority; p = 0.2496, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -6.3
Statistical Analysis 4: Comparison: Baloxavir Marboxil vs Oseltamivir; Sore Throat; Test type: Superiority; p = 0.2963, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = 0.9
Statistical Analysis 5: Comparison: Baloxavir Marboxil vs Placebo; Headache; Test type: Superiority; p = 0.0390, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -10.6
Statistical Analysis 6: Comparison: Baloxavir Marboxil vs Oseltamivir; Headache; Test type: Superiority; p = 0.7877, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = 2.0
Statistical Analysis 7: Comparison: Baloxavir Marboxil vs Placebo; Nasal Congestion; Test type: Superiority; p = 0.0017, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -12.1
Statistical Analysis 8: Comparison: Baloxavir Marboxil vs Oseltamivir; Nasal Congestion; Test type: Superiority; p = 0.8119, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = 1.5
Statistical Analysis 9: Comparison: Baloxavir Marboxil vs Placebo; Feverishness or Chills; Test type: Superiority; p = 0.0070, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -3.6
Statistical Analysis 10: Comparison: Baloxavir Marboxil vs Oseltamivir; Feverishness or Chills; Test type: Superiority; p = 0.9191, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -0.7
Statistical Analysis 11: Comparison: Baloxavir Marboxil vs Placebo; Muscle or Joint Pain; Test type: Superiority; p = 0.0232, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -7.7
Statistical Analysis 12: Comparison: Baloxavir Marboxil vs Oseltamivir; Muscle or Joint Pain; Test type: Superiority; p = 0.5436, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = 4.0
Statistical Analysis 13: Comparison: Baloxavir Marboxil vs Placebo; Fatigue; Test type: Superiority; p = 0.0207, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -7.5
Statistical Analysis 14: Comparison: Baloxavir Marboxil vs Oseltamivir; Fatigue; Test type: Superiority; p = 0.3710, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -1.9

18. Secondary Outcome: Time to Return to Preinfluenza Health Status
Description: Participants were asked to record their preinfluenza health status on a scale from 0 (worst possible health) to 10 (normal health [for someone your age and condition]), and their health status at baseline and every day after initiation of study treatment on the same scale. Return to preinfluenza health status was defined as time from the initiation of the study treatment to the first time when the health status score was equal to or higher than the preinfluenza health status score.
  Time to return to preinfluenza health status was analyzed using KM methods; participants with a smaller number on the scale for health status by the last observation time point were censored at that time point.
Time Frame: Baseline to Day 14
Population: Participants in the intention-to-treat infected population whose health status score at baseline was lower than the preinfluenza health status score and with available time to return to preinfluenza health status data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 274 | 274 | 286
hours | 126.4 [104.6 to 153.4] | 149.8 [124.7 to 175.7] | 126.9 [104.9 to 152.7]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.4634, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -23.4
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.6386, Generalized Wilcoxon test — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05; [statistical method as in outcome 1, analysis 1]; Median Difference = -0.6

19. Secondary Outcome: Percentage of Participants Requiring Systemic Antibiotics for Infections Secondary to Influenza Infection
Description: The percentage of participants who received systemic antibiotics for any of the predefined complications (sinusitis, otitis media, bronchitis and pneumonia).
Time Frame: Day 2 to Day 22
Population: Intention-to-treat infected population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 388 | 386 | 389
percentage of participants | 3.4 [1.8 to 5.7] | 7.5 [5.1 to 10.6] | 3.9 [2.2 to 6.3]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Test type: Superiority; p = 0.0112, Fisher Exact — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Test type: Superiority; p = 0.8478, Fisher Exact — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05

20. Secondary Outcome: Percentage of Participants With Influenza-related Complications
Description: Defined as the percentage of patients who experience each influenza-related complication (hospitalization, death, sinusitis, otitis media, bronchitis, and radiologically-confirmed pneumonia) as an adverse event after the initiation of study treatment.
Time Frame: Day 1 to Day 22
Population: Intention-to-treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 388 | 386 | 389
percentage of participants
  Any Complications | 2.8 [1.4 to 5.0] | 10.4 [7.5 to 13.8] | 4.6 [2.8 to 7.2]
  Death | 0.0 [0.0 to 0.9] | 0.0 [0.0 to 1.0] | 0.3 [0.0 to 1.4]
  Hospitalization | 0.8 [0.2 to 2.2] | 1.3 [0.4 to 3.0] | 1.0 [0.3 to 2.6]
  Sinusitis | 0.3 [0.0 to 1.4] | 2.1 [0.9 to 4.0] | 0.5 [0.1 to 1.8]
  Otitis media | 0.0 [0.0 to 0.9] | 0.8 [0.2 to 2.3] | 0.3 [0.0 to 1.4]
  Bronchitis | 1.8 [0.7 to 3.7] | 6.0 [3.8 to 8.8] | 2.3 [1.1 to 4.3]
  Pneumonia | 0.0 [0.0 to 0.9] | 0.8 [0.2 to 2.3] | 0.5 [0.1 to 1.8]
Statistical Analysis 1: Comparison: Baloxavir Marboxil vs Placebo; Any Complications; Test type: Superiority; p < 0.0001, Fisher Exact — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05
Statistical Analysis 2: Comparison: Baloxavir Marboxil vs Oseltamivir; Any Complications; Test type: Superiority; p = 0.2558, Fisher Exact — The p value was not adjusted for multiplicity, testing was conducted at the two-sided significance level of 0.05

21. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: From first dose of study drug to Day 22
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
Number analyzed (Participants) | 730 | 727 | 721
percentage of participants
  Any adverse event (AE) | 25.1 | 29.7 | 28.0
  Fatal adverse events | 0.0 | 0.0 | 0.1
  Serious adverse events | 0.7 | 1.2 | 1.1
  AEs leading to withdrawal of study drug | 0.7 | 0.7 | 0.6
  Treatment-related adverse events (TRAEs) | 5.6 | 8.3 | 7.9
  Fatal treatment-related adverse events | 0.0 | 0.0 | 0.0
  Treatment-related serious adverse events | 0.0 | 0.3 | 0.3
  TRAEs leading to withdrawal of study drug | 0.3 | 0.3 | 0.4

ADVERSE EVENTS:
Time Frame: All-cause mortality data are reported from Day 1 though Day 22. Adverse events are reported from the first dose of study drug through Day 22 (i.e. treatment-emergent adverse events).
Description: One participant randomized to placebo and one participant randomized to oseltamivir received baloxavir marboxil in error, and are counted in the baloxavir marboxil, treatment group for safety analyses.
  One participant died after a myocardial infarction that occurred prior to receiving any study drug; although this death is included in the all-cause mortality table this death was not considered treatment-emergent.
Arm/Group | Baloxavir Marboxil | Placebo | Oseltamivir
All-Cause Mortality (participants affected / at risk) | 1/730 | 0/727 | 1/721
Serious Adverse Events (participants affected / at risk) | 5/730 | 9/727 | 8/721
Other Adverse Events (participants affected / at risk) | 70/730 | 92/727 | 90/721
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baloxavir Marboxil (N=730) | Placebo (N=727) | Oseltamivir (N=721)
Pneumonia (Infections and infestations) | 1 | 1 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Arachnoid cyst (Nervous system disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Baloxavir Marboxil (N=730) | Placebo (N=727) | Oseltamivir (N=721)
Bronchitis (Infections and infestations) | 21 | 33 | 30
Sinusitis (Infections and infestations) | 14 | 21 | 22
Diarrhoea (Gastrointestinal disorders) | 20 | 21 | 23
Nausea (Gastrointestinal disorders) | 20 | 28 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT02949011/SAP_001.pdf
  • Study Protocol (2016-10-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT02949011/Prot_002.pdf